CLINICAL TRIAL: NCT04451382
Title: Treatment of Refractory Overactive Bladder (OAB) With OnabotulinumtoxinA vs. PTNS: TROOP Trial
Brief Title: PTNS vs Botox of Refractory OAB
Acronym: TROOP
Status: Terminated | Type: Observational
Why Stopped: Low recruitment
Sponsor: Medstar Health Research Institute (Other)
Collaborators: University of Michigan (Other); Methodist Urology Associates, Houston, Texas (Unknown); Columbia University (Other); University of New Mexico (Other)
Responsible Party: Principal Investigator, Robert Gutman, MD, Medstar Health Research Institute
Other Study IDs: 2014-277
Record Dates: First submitted 2015-10-31; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Overactive Bladder (OAB)
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OnabotulinumtoxinA (BoNTA): DRUG: OnabotulinumtoxinA (BoNTA) is an injection into the bladder which blocks the presynaptic release of acetylcholine. BoNTA was approved for the treatment of OAB by the FDA in 2013.
  Interventions: Biological: OnabotulinumtoxinA (BoNTA)
- Percutaneous tibial nerve stimulation (PTNS): DEVICE: PTNS involves needle stimulation of the posterior tibial nerve and is typically performed with weekly 30 minute sessions for a 12 week treatment course.
  Interventions: Procedure: Percutaneous tibial nerve stimulation (PTNS)

INTERVENTIONS:
Biological: OnabotulinumtoxinA (BoNTA)
  Other Names: Botox
  Groups: OnabotulinumtoxinA (BoNTA)
Procedure: Percutaneous tibial nerve stimulation (PTNS)
  Groups: Percutaneous tibial nerve stimulation (PTNS)

SUMMARY:
This is a prospective cohort study of women with overactive bladder OAB (dry or wet) who have failed 2 prior treatments, including behavioral modification, pelvic floor physical therapy, and/or OAB medication (anticholinergics or mirabegron), and have chosen either OnabotulinumtoxinA (BTX) injection or percutaneous tibial nerve stimulation (PTNS) as their next treatment. OAB-dry refers to patients with OAB who do not have urge urinary incontinence; OAB-wet refers to patients with OAB and urge urinary incontinence. Eligible patients will be approached for study participation after they have decided to proceed with BTX or PTNS.

DETAILED DESCRIPTION:
Prior to initiation of BTX or PTNS, patients will undergo a standardized evaluation including urodynamics study (UDS) if not previously done in the past year and pelvic organ prolapse quantification (POPq) exam if not previously done in past 6 months. Subjects will also complete quality of life questionnaires and 3-day voiding diary prior to initial treatment. Follow up questionnaires will be completed at 3 months either in office, if patient has a routine visit scheduled with provider and questionnaires can be completed at that visit or questionnaires will be mailed with return postage for participant to mail completed questionnaires back.

ELIGIBILITY:
Inclusion Criteria:

1. Women with refractory OAB (dry or wet)
2. OAB will be defined by a positive response and bother of "somewhat, quite a bit, a great deal, or a very great deal" to question #3 or #8 on the OAB-q (see appendix B) regarding urinary urgency and urgency incontinence.
3. Refractory will be defined as failure of 2 prior treatments, including behavioral modification, pelvic floor physical therapy, and OAB medication (anticholinergics or mirabegron). Trial of 2 medications that did not improve symptoms after 2 weeks or could not be tolerated due to side effects will constitute 2 treatment failures.
4. Women with mixed urinary incontinence that is urge predominant will also be included.
5. Age ≥ 18 years
6. English speaking
7. Available for 1 year follow-up
8. Able to complete study questionnaires

Exclusion Criteria:

1. Neurologic disease known to cause OAB including, but not limited to, Multiple sclerosis, Parkinson's disease, and Spinal Cord Injury.
2. Pregnancy by self-report or pregnancy test
3. Contraindication to PTNS and/or BTX

   * PTNS: Pacemaker
   * BTX: myasthenia gravis, allergy to BTX, urinary retention (post void residual >200cc)
4. Planned surgery for pelvic floor disorder during the study period
5. Prior treatment with BTX, PTNS, or sacral nerve stimulation (SNS) for refractory OAB/urinary urge incontinence (UUI)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with refractory OAB (dry or wet) who have failed 2 prior treatments, including behavioral modification, pelvic floor physical therapy, and/or OAB medication (antimuscarinics or mirabegron), and have chosen either BTX or PTNS as their next treatment.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Difference in patient global impression of improvement score between PTNS and BTX groups | 3 month
  The Patient Global Impression of Improvement (PGI-I) is a single question that asks a patient to rate her urinary symptom response to treatment on a 7-point Likert scaleis a validated questionnaire for assessment of the impact of OAB on patient's lives.
Change in quality of life between PTNS and BTX groups | 3 month
  The minimally important difference (MID) for change in SSS is 10 points. We compare the change in SS score between the PTNS and Botox groups at 3 months.

SECONDARY OUTCOMES:
Change in individual question scores on OAB-q questionnaire | 3
  The OAB-q consists of 33 items: an 8-item symptom bother scale (SS) and a 25-item health-related quality of life (HRQL) scale. Higher scores on HRQL scale represent better quality of life and lower scores on SSS is indicative of less bother.
Change in urinary symptom severity | 3
  Tools used: Urogenital Distress Inventory short form (UDI-6) is a validated questionnaires used to assess urinary symptoms. We will compare change in scores between the 2 groups

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Columbia University, New York, New York